CLINICAL TRIAL: NCT02492126
Title: Chronic Cough and Reflux: Is Esophageal Motility the Key?
Brief Title: Esophageal Motility in Reflux Induced Cough
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Principal Investigator, Kenneth R. DeVault, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 15-002020
Record Dates: First submitted 2015-07-02; First posted 2015-07-08 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Cough
Keywords: Chronic Cough; Gastroesophageal Reflux; Esophageal Motility; Cough Sensitivity
MeSH Terms: conditions — Cough; Chronic Cough; Gastroesophageal Reflux | interventions — Citric Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Cough: Subjects with chronic cough will undergo cough reflex sensitivity testing to citric acid. The dose, starting at 0.03 mol/L citric acid will be administered as single breath inhalations using flow-limited calibrated pots and a dosimeter with 3 placebo inhalations of normal saline randomly interspersed. Following each inhalation, the number of coughs in the subsequent 15 seconds will be counted and recorded. The challenge will be terminated once the citric acid has induced 5 or more coughs.
  Interventions: Other: Citric Acid

INTERVENTIONS:
Other: Citric Acid — Subjects will undergo cough reflex sensitivity testing to citric acid.

SUMMARY:
To determine whether contraction abnormalities in the esophagus plays a role in gastroesophageal reflux induced cough, and thus cough severity in patients with chronic cough.

ELIGIBILITY:
Inclusion criteria:

1. Adult patients (ages 18-75 years old)
2. Cough for more than 8 weeks
3. Additional clinical evaluation of cough including a complete pulmonary function test with methacholine challenge and a high resolution CT scan of the chest.
4. Ability to understand the purpose and nature of the study
5. Willingness to participate and provide consent form

Exclusion criteria:

1. Actively smoke in the preceding 6 months.
2. Recent respiratory tract infection (<4 weeks).
3. Drink above the recommended safe alcohol limit (21 units per week).
4. History of respiratory or gastrointestinal malignancies.
5. Previous gastrointestinal surgery (excluding minor surgeries, such as cholecystectomy, appendectomy).
6. Subjects with established and significant cardiac, pulmonary, or neurological disorders as deemed by the clinician or study personnel
7. Use of angiotensin converting enzyme inhibitors
8. Use of H2 blockers or proton pump inhibitors in the seven days prior to reflux testing (impedance/pH), or inability to withhold such medications for the duration of the study
9. Women of childbearing potential, using adequate birth control. Adequate birth control includes: (i) hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants; (ii) barrier methods (such as, a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm); (iii) intrauterine device (IUD); or (iv) abstinence (no sex). Adequate birth control must be maintained for the duration of the study. Women not using adequate birth control will be excluded from the study, as funding for the pregnancy tests was not included in the small grant awarded for this study.
10. Nursing mothers will be excluded.
11. Persons with allergies to citrus will be excluded.
12. Inability to understand the purpose and nature of the study
13. Unwillingness to participate and provide consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic cough patients
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with reflux related cough | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth DeVault, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials